CLINICAL TRIAL: NCT01143168
Title: A Pilot Study on Transplantation Therapy Using Autologous Bone Marrow Mononuclear Cells and Umbilical Cord Mesenchymal Stem Cells in Patients With Type 1 Diabetes Mellitus
Brief Title: Stem Cell Therapy for Type 1 Diabetes Mellitus
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cellonis Biotechnology Co. Ltd. (Industry)
Responsible Party: Cellonis Biotechnology Co. Ltd., Others
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cellonis-CR-1.3
Record Dates: First submitted 2010-06-10; First posted 2010-06-14 (Estimated); Last update posted 2010-06-14 (Estimated); Status verified 2010-06

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: stem cells;; diabetes mellitus;; treatment.
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: autologous bone marrow mononuclear cells and umbilical cord mesenchymal stem cells — First Transplantation: after finishing all required examines according to protocol on Day 0, ABM-MNCs + UCMSCs are transplanted through pancreas artery percutaneously; Second Transplantation: after finishing all required examines on Day 7±1, BM-MNCs UCMSCs are transplanted intravenously; Third Transplantation: after finishing all required examines on Day 14±2, BM-MNCs + UCMSCs are transplanted intravenously.

SUMMARY:
The purpose of this study is to evaluate the feasibility, efficacy and safety of transplantation therapy using bone marrow mononuclear cells and umbilical cord mesenchymal stem cells for patients with type 1 diabetes mellitus

DETAILED DESCRIPTION:
To evaluate the feasibility, safety and efficacy of transplantation using autologous bone marrow mononuclear cells and umbilical cord mesenchymal stem cells in patients with type 1 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Free will taking part in the study and ability to provide written informed consent.
2. Confirmed diagnosis of type I diabetes for at least 2 years
3. Insulin-dependent.
4. Age 18-50 years, Male/Female.
5. FBG≥7.0 mmol/L, and HbAc1≥7％.
6. Not pregnant or nursing.
7. Negative pregnancy test.
8. Fertile patients will use effective contraception.

Exclusion Criteria:

1. Presence of acute diabetic complications in the acute stage as recent myocardial infarction, recent cerebral vascular accident (CVA) or acute renal failure.
2. Severe concurrent medical condition (e.g. lung disease, or hematopoietic dysfunction, or liver dysfunction).
3. Active infection requiring treatment.
4. Known immunosuppressive disease, e.g. HIV infection, or hepatitis B or C infection.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-08 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Rate of reducing exogenous insulin requirement; Hemoglobin A1c; Fast blood glucose (FBG) and postmeal blood glucose (PBG); C-peptide levels. | 1 year
  Rate of reducing exogenous insulin requirement compared with baseline. Hemoglobin A1c. Fast blood glucose (FBG) and postmeal blood glucose (PBG). C-peptide levels.

SECONDARY OUTCOMES:
Serious adverse event frequency and severity | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shi X Y, M.D., Principal Investigator — Armed Police General Hospital, P. R. China
Locations (1):
- Armed Police General Hospital, P. R. China, Beijing, China